CLINICAL TRIAL: NCT02886013
Title: FTO rs9939609 and PPARy rs1801282 Polymorphisms in Mexican Adolescents With Overweight and Obesity at High Risk for Developing Diabetes
Brief Title: FTO rs9939609 and PPARy rs1801282 Polymorphisms in Mexican Adolescents
Status: Completed | Type: Observational
Sponsor: Asociación Científica Latina A.C. (Other)
Responsible Party: Principal Investigator, Dr. Hugo Mendieta Zerón, Director, Asociación Científica Latina A.C.
Other Study IDs: 2016-03
Record Dates: First submitted 2016-08-21; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: prevalence
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 mL of venous blood (Vacutainer tubes) were taken in fasting. A sample remained frozen at -70°C (900 series Thermo Scientific) until DNA extraction.
  Genotyping DNA extraction was performed in the Magna Pure LC 2.0 Instrument (Roche, Germany) using the MagNA Pure LC DNA Isolation Kit 1 (Roche, Germany).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mexican adolescents: Students without known disease, between 14 and 18 years from the "Lic. Adolfo Lopez Mateos" Preparatory school of the Autonomous University of the State of Mexico (UAEMex).

SUMMARY:
Background and Aims: The presence of the FTO rs9939609 and PPARy rs1801282 polymorphisms suggests changes in energy metabolism; this variation may be responsible for the development of various diseases including obesity. The aim of this study was to identify the presence of these polymorphisms in Mexican adolescents with overweight and obesity at high risk for developing diabetes. Methods and Results: This was a descriptive cross-sectional study, where 71 healthy adolescents (average age of 16) were included. Anthropometric measurements, Body mass index, as well as the determination of glucose, insulin and HOMA index were calculated from all the patients. The FTO rs9939609 and PPARy rs1801282 polymorphisms were determined by real-time PCR.

DETAILED DESCRIPTION:
Study Population Students without known disease, between 14 and 18 years from the "Lic. Adolfo Lopez Mateos" Preparatory school of the Autonomous University of the State of Mexico (UAEMex), were invited to participate.

Anthropometry The body mass index (BMI) was calculated as weight (kg) divided by height (m) squared with conventional stadiometer; dividing the results in normal, overweight and obesity according to the classification of the World Health Organization (WHO), specifically for adolescents by gender and age.

Laboratory 3 mL of venous blood (Vacutainer tubes) were taken in fasting. The concentration of glucose, total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides were determined by enzymatic methods (Randox Laboratories Ltd, County Antrim, UK); whereas leptin and adiponectin concentrations were determined by the immunosorbent assay (ELISA) (Invitrogen MR Frederyck MD USA). A sample remained frozen at -70°C (900 series Thermo Scientific) until DNA extraction.

Genotyping DNA extraction was performed in the Magna Pure LC 2.0 Instrument (Roche, Germany) using the MagNA Pure LC DNA Isolation Kit 1 (Roche, Germany). After extraction, the DNA was quantified using a NanoPhotometer (Implen GmbH, Germany), reporting concentration (μg/ml) and purity (260/280 absorbance). Genotyping was performed by polymerase chain reaction (PCR) Life express thermal cycler (Bioer, China). The primers and conditions for each polymorphism are listed in Table 1.

The oligonucleotides were designed using the Primer Quest web tool (Integrated DNA Technologies, Inc., CA, USA) and synthesized at the Synthesis and DNA Sequencing Unit of the National Autonomous University of Mexico (UNAM) Institute of Biotechnology (Cuernavaca, Morelos, Mexico). A search was performed in BLAST to verify the correct hybridization. The final products were visualized in 2% agarose gels, stained with ethidium bromide, and visualized under an UV transilluminator (Gel Logic 212 Pro, Carestream, USA). To confirm the detection of polymorphisms sequencing was performed at the National Institute of Genomic Medicine (INMEGEN), Mexico City.

ELIGIBILITY:
Inclusion Criteria:

* Students without known disease, between 14 and 18 years from the "Lic. Adolfo Lopez Mateos" Preparatory school of the Autonomous University of the State of Mexico (UAEMex).

Exclusion Criteria:

* Those with a history of smoking, pregnancy or diagnosed with a chronic diseases.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mexican adolescents with overweight and obesity at high risk for developing diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of the FTO rs9939609 and PPARy rs1801282 polymorphisms. | up to 24 months.
  The aim of this study was to identify the presence of these polymorphisms in Mexican adolescents with overweight and obesity at high risk for developing diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: María del Socorro Camarillo Romero, PhD., Study Chair — Autonomous University of the State of Mexico

IPD SHARING:
Plan to Share IPD: No